CLINICAL TRIAL: NCT03686254
Title: The Effect and Safety on Unresectable CRLM From RFA in Combination With Second-line Chemotherapy and Bevacizumab Compared With the Combination of Second-line Chemotherapy and Bevacizumab: a Randomized and Controlled Clinical Trial
Brief Title: The Effects of RFA in Combination With Second-line Chemotherapy and Bevacizumab on Unresectable CRLM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Wangjun Liao, Chief of Oncology Department, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2016ZD014
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Neoplasms Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — Radiofrequency Ablation; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control Arm (Active Comparator): bevacizumab and second-line chemotherapy
  Interventions: Drug: Bevacizumab and second-line chemotherapy
- The experimental Arm (Experimental): RFA, bevacizumab and second-line chemotherapy
  Interventions: Combination Product: RFA, bevacizumab and second-line chemotherapy

INTERVENTIONS:
Combination Product: RFA, bevacizumab and second-line chemotherapy — Navigated by CT-ultrasound merged images, RFA is taken in the experimental arm at the first day of the first cycle during the second-line therapy. Bevacizumab is given to patients in all arms every 2 weeks (5mg/kg) or 3 weeks (7.5mg/kg), intravenous drip(VD). The second-line chemotherapies include FOLFIRI [Irinotecan 180 mg/m2 D1+Calcium folinatc 400 mg/m2 or Calcium Levofolinate 200 mg/m2 D1+5-FU 400 mg/m2 D1, 2400 mg/m2 D1-2(46-48h), q2W] or irinotecan monotherapy (125 mg/m2 D1, 8, q3W or 180 mg/m2 D1, q2W), mFOLFOX6 [Oxaliplatin 85 mg/m2 D1+Calcium folinatc 400 mg/m2 or Calcium Levofolinate 200 mg/m2 D1+5-FU 400 mg/m2 D1, 2400 mg/m2 D1-2(46-48h), q2W] or CapeOX (Oxaliplatin 130 mg/m2 D1+Capecitabine 1000 mg/m2 Bid D1-14, q3W)，or irinotecan+oxaliplatin (Oxaliplatin 85 mg/m2 D1+Irinotecan 200 mg/m2 D1, q3W). Among these strategies, the treatment cycle of FOLFIRI, irinotecan monotherapy and mFOLFOX6 is two weeks, while three weeks in CapeOX and irinotecan + oxaliplatin.
  Arms: The experimental Arm
Drug: Bevacizumab and second-line chemotherapy — Bevacizumab is given to patients in all arms every 2 weeks (5mg/kg) or 3 weeks (7.5mg/kg), intravenous drip(VD). The second-line chemotherapies include FOLFIRI [Irinotecan 180 mg/m2 D1+Calcium folinatc 400 mg/m2 or Calcium Levofolinate 200 mg/m2 D1+5-FU 400 mg/m2 D1, 2400 mg/m2 D1-2(46-48h), q2W] or irinotecan monotherapy (125 mg/m2 D1, 8, q3W or 180 mg/m2 D1, q2W), mFOLFOX6 [Oxaliplatin 85 mg/m2 D1+Calcium folinatc 400 mg/m2 or Calcium Levofolinate 200 mg/m2 D1+5-FU 400 mg/m2 D1, 2400 mg/m2 D1-2(46-48h), q2W] or CapeOX (Oxaliplatin 130 mg/m2 D1+Capecitabine 1000 mg/m2 Bid D1-14, q3W)，or irinotecan+oxaliplatin (Oxaliplatin 85 mg/m2 D1+Irinotecan 200 mg/m2 D1, q3W). Among these strategies, the treatment cycle of FOLFIRI, irinotecan monotherapy and mFOLFOX6 is two weeks, while three weeks in CapeOX and irinotecan + oxaliplatin.
  Arms: The control Arm

SUMMARY:
Basing on the strong evidence from former researches, patients with CRLM can benefit from the treatment of bevacizumab combined with sencond-line chemotherapy. Recently, although with the popularization of RFA, the role that RFA plays in the long term survival of patients with metastatic colorectal cancer (CRC) is still confused. In this designed, randomized, controlled, prospective, and open clinical trial, the effectiveness of RFA combined with second-line chemotherapy + bevacizumab on unresectable CRLM is going to be evaluated compared with that of second-line chemotherapy + bevacizumab. After screened by inclusion and exclusion criteria, the eligible subjects will be randomly allocated into the experimental group-with the treatment of RFA + second-line chemotherapy + bevacizumab and control group-with the treatment of second-line chemotherapy + bevacizumab equally.

DETAILED DESCRIPTION:
As a leading cause of death around the world, the mobility and mortality of CRC also increase in china with aging. Currently, distant organ metastasis, most commonly appearing in liver, diminishes the life expectancy in more than 50% of CRC patients. Surgical resection of the tumor primaries and metastases has been the first choice of patients with CRLM with five-year survival rate of 44.2%. With only 25% resectable CRLM, however, most patients lose the operation chance at diagnosis.

In the past two decades, RFA in CRLM treatment has been gradually approved and showed great value in clinic. According to some retrospective researches, for small metastases, the effectiveness of RFA is not inferior to surgery. However, what really makes sense is to ensure if patients with unresectable metastases could benefit from RFA. The results from some former researches and CLOCC study in 2017 noticeably reflected that RFA enabled to prolong the survival significantly in unresectable CRLM patients, which determined its essential role in clinical application.

As a humanized monoclonal antibody against vascular endothelial growth factor (VEGF), bevacizumab shows great potential in tumor therapy: pruning the tumor vessels rapidly by blocking VEGF signaling pathway; straightening and normalizing tumor vessels which ensure the effective perfusion of chemotherapeutics. In addition, depending on durable angiogenesis inhibition, bevacizumab restrains tumor growth and metastasis. To date, bevacizumab combined with chemotherapy is approved in metastatic CRC treatment.

For long term survival, patients with CRLM can benefit from bevacizumab combined with sencond-line chemotherapy basing on the strong evidence from above researches. While the role that RFA plays in this therapeutic regimen is still confused. In this designed clinical trial, the main purpose is to evaluate the effectiveness of RFA combined with second-line chemotherapy + bevacizumab on CRLM patients plans, which is expected to polish up the clinical treatment approaches.

This study is a randomized, controlled, prospective, open, and two-center clinical experiment for patients with metastatic CRC. After screened by inclusion and exclusion criteria, the eligible subjects will be randomly allocated into the experimental group and control group equally. Liver biopsy or specimens of liver metastases are required in all eligible patients for the second pathologic diagnosis by pathology department in Nanfang hospital, Southern Medical University.

Supported by Logrank test in PASS II software, this study will compare the survival differences between experimental and control group. In CLOCC study, the ratio between hazard ratio (HR) of chemotherapy bevacizumab combined with RFA and that of chemotherapy bevacizumab was 0.58. Considering that the subjects in this study are after second-line therapy and extrahepatic metastases are allowed, so the HR will supposedly achieve 0.62. In addition, with the four stratified blocks and 5% expulsion rate in both experimental and control groups, 80 subjects in each group (total 160 subjects) are needed to detect the difference with 80% confidence at the a=0.05 (bilateral) significant level.

In control group, subjects are treated with bevacizumab + second-line chemotherapy, while treated with RFA + bevacizumab + second-line chemotherapy in experimental group. The detailed descriptions of these interventions are as follow. Bevacizumab is given to patients in all arms every 2 weeks (5mg/kg) or 3 weeks (7.5mg/kg), intravenous drip(VD). The second-line chemotherapies depending on the judgement of researchers and the wills of subjects include FOLFIRI [Irinotecan 180 mg/m2 D1+Calcium folinatc 400 mg/m2 or Calcium Levofolinate 200 mg/m2 D1+5-FU 400 mg/m2 D1, 2400 mg/m2 D1-2(46-48h), q2W] or irinotecan monotherapy (125 mg/m2 D1, 8, q3W or 180 mg/m2 D1, q2W) with the historical first-line treatment of oxaliplatin but not irinotecan, mFOLFOX6 [Oxaliplatin 85 mg/m2 D1+Calcium folinatc 400 mg/m2 or Calcium Levofolinate 200 mg/m2 D1+5-FU 400 mg/m2 D1, 2400 mg/m2 D1-2(46-48h), q2W] or CapeOX (Oxaliplatin 130 mg/m2 D1+Capecitabine 1000 mg/m2 Bid D1-14, q3W) with the historical first-line treatment of irinotecan but not oxaliplatin, and mFOLFOX6, CapeOX, FOLFIRI, irinotecan monotherapy or irinotecan+oxaliplatin (Oxaliplatin 85 mg/m2 D1+Irinotecan 200 mg/m2 D1, q3W) with the historical first-line treatment of fluorouracil but not oxaliplatin and irinotecan. Among these strategies, the treatment cycle of FOLFIRI, irinotecan monotherapy and mFOLFOX6 is two weeks, while three weeks in CapeOX and irinotecan + oxaliplatin. Navigated by CT-ultrasound merged images, RFA is taken in the experimental arm at the first day of the first cycle during the second-line therapy. The initial power is 30w and increases 20w per minute until 90w is reached. Then the operation will last for 15 minutes or until the power fall to 0w. If any severe unfit or abnormal vital signs occur in subjects during the process and cannot be improved by symptomatic treatment, RFA should be stopped immediately. After ensuring that the ablation area assessed by the hyperechoic area in ultrasound has reached the intended target, the operation finishes successfully and postoperative observation (including pulse, breath, and blood pressure etc.) is needed in all experimental patients. To make the residual volumes of metastases as small as possible, repeated RFA can be operated within 1 week after initial RFA treatment if the criteria of normal coagulation function, platelets (PLT) 80/L and neutrophils 1.5/L, and RFA related adverse events grade 1 are satisfied, but at most 3 times.

Tumor burden will be evaluated by imaging according to RECIST 1.1. For the assessment of baseline level and at the first day ( 3 days) of the second cycle, PET-CT is designated. While the subsequent method-enhanced CT or MRI is determined by researchers. Thoracic, abdominal and pelvic examinations are involved at each assessment. And the evaluation should be taken every 2 months ( 7 days) until progression or deaths occur. Baseline assessment refers to whole body PET-CT, and additional head CT/MRI or bone scanning are required if suspected brain or osseous metastases exist.

The safety will be evaluated through the analysis of adverse events (AE), severe adverse events (SAE) and laboratory abnormalities, especially the specific events-hemorrhage and elevated transaminase. The observational parameters include the type, incidence, severity, time, correlation, risk factors, measurements and outcomes. The severity of every AE will be classified into 5 grades according to National Cancer Institute (NCI-CTCAE), v 4.03. Main researcher will be responsible for the documentation of AE and SAE.

The study will conduct at 24-month baseline and 36-month follow-up, and the anticipated duration is 5 years.

ELIGIBILITY:
Inclusion Criteria:

1.CRLM patients with histopathological diagnosis. 2.Tumor progression after first-line therapy or intolerable adverse events occur;

1. The first-line therapy should be the standard regimen recommended by NCCN guideline.
2. Tumor progression indicates: progression occurs during the process or within three months after the final treatment of first-line therapy; progression occurs during the period of adjunctive therapy/neoadjuvant therapy or within six months after adjunctive therapy finished.
3. Prior treatment with bevacizumab or cetuximab is allowed. 3.Aged between 16-80 years old (16 and 80 years old are included), with no limitation of gender; 4.ECOG scores 0-1; 5.At least one measurable liver metastasis according to RECIST 1.1 criteria; 6.The liver metastasis is no larger than 50% of total liver lesions; 7.Determined as unresectable liver metastasis by the multidisciplinary team consisting of liver surgeons and medical oncologists;

1)R0 resection cannot be operated on liver metastases. 2)Hepatic artery or the branches of portal vein is invaded. 3)The three main hepatic veins are surrounded by liver metastases. 4)Extrahepatic metastases coexist. 8.Life expectancy is above three months; 9.With full appreciation, voluntary and a signed informed consent; 10.Vital organs with normal function:

1. Routine blood test: hemoglobin (HGB) 85g/L, platelet (PLT) 80/L, and neutrophils 1.5/L;
2. Normal coagulation function originally or after treatment (if exceeding reference level, whether it is still within normal range should be determined by researchers);
3. Total bilirubin(BIL) is 1.5 times higher than the upper normal limit, alanine aminotransferase (ALT) and aspartic transaminase (AST) are 5 times higher than the upper normal limit;
4. Urine protein ranges from - to +, and serum creatinine 1.5×ULN; 11.Negative pregnancy test results in women of childbearing age (7 days before RFA treatment), and effective contraceptive measures must be adopted until 6 m after the last treatment.

Exclusion Criteria:

1. Prior treatment with other clinically experimental drugs, systemic chemotherapy, immunotherapy or targeted therapy within 2 weeks before this trial;
2. Prior treatment on liver metastases with radiotherapy, hepatic arterial infusion chemotherapy, transcatheter hepatic arterial chemoembolization, cryoablation, microwave ablation or RFA within 2 weeks before this trial;
3. Abnormal coagulation function and with hemorrhagic tendency;
4. Damaged or infectious skin in the puncture or electrode sticking area;
5. Complicated by active hepatitis or hepatic failure;
6. Complicated by severe hypertension or hypertensive crisis (systolic pressure 180 mmHg and/or diastolic pressure 110 mmHg in a resting state);
7. Impaired cardiac function, manifested as left ventricular ejection fraction 50%, severe arrhythmia, unstable angina, history of myocardial infarction within 1 year before this trial, or congestive heart-failure in NYHA class III or IV;
8. History of stroke within 6 months;
9. History of other malignancies except for colorectal cancer within 5 years;
10. Abnormal medical or psychologic status that may hamper the ongoing trial or signing an informed consent;
11. No or limited legal capacity;
12. Pregnant or breast-feeding women;
13. Combined acute infection or human immunodeficiency virus (HIV) infection;
14. With contradictions for bevacizumab; 1)History of severe hemorrhage or hemoptysis 1 month before this trial 2)Urine protein 2+, and 24-hour urinary protein quantitative 2g 3)Allergy to bevacizumab or any active ingredients 4)Patients with surgery, major trauma or fracture within 4 weeks 5)Unhealed wounds, intestinal stomas or peptic ulcer
15. Treated with other experimental antineoplastic drugs.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS), Month | From the date of randomization until the date of death due to any cause, assessed up to 36 months

SECONDARY OUTCOMES:
Progress free survival (PFS), Month | From the date of randomization until the date of first documented tumor progression or date of death before progression due to any cause, assessed up to 36 months
Time to progression (TTP), Month | From the date of randomization until the date of first documented tumor progression, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Wangjun Liao, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hur H, Ko YT, Min BS, Kim KS, Choi JS, Sohn SK, Cho CH, Ko HK, Lee JT, Kim NK. Comparative study of resection and radiofrequency ablation in the treatment of solitary colorectal liver metastases. Am J Surg. 2009 Jun;197(6):728-36. doi: 10.1016/j.amjsurg.2008.04.013. Epub 2008 Sep 11. PMID 18789428
- [Background] Giantonio BJ, Catalano PJ, Meropol NJ, O'Dwyer PJ, Mitchell EP, Alberts SR, Schwartz MA, Benson AB 3rd; Eastern Cooperative Oncology Group Study E3200. Bevacizumab in combination with oxaliplatin, fluorouracil, and leucovorin (FOLFOX4) for previously treated metastatic colorectal cancer: results from the Eastern Cooperative Oncology Group Study E3200. J Clin Oncol. 2007 Apr 20;25(12):1539-44. doi: 10.1200/JCO.2006.09.6305. PMID 17442997
- [Result] Ruers T, Van Coevorden F, Punt CJ, Pierie JE, Borel-Rinkes I, Ledermann JA, Poston G, Bechstein W, Lentz MA, Mauer M, Folprecht G, Van Cutsem E, Ducreux M, Nordlinger B; European Organisation for Research and Treatment of Cancer (EORTC); Gastro-Intestinal Tract Cancer Group; Arbeitsgruppe Lebermetastasen und tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); National Cancer Research Institute Colorectal Clinical Study Group (NCRI CCSG). Local Treatment of Unresectable Colorectal Liver Metastases: Results of a Randomized Phase II Trial. J Natl Cancer Inst. 2017 Sep 1;109(9):djx015. doi: 10.1093/jnci/djx015. PMID 28376151